CLINICAL TRIAL: NCT00963508
Title: A Multi-Center Phase III Study to Evaluate Malathion Gel 0.5% Formulation, for the Control of Head Lice in Pediatric Subjects and Adult Subjects With Pediculosis Capitis
Brief Title: Efficacy, Safety and Tolerability of a Novel Malathion Formulation in Patients 2 Years and Older With Head Lice
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MALG-0816
Record Dates: First submitted 2009-08-14; First posted 2009-08-21 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-05

CONDITIONS: Pediculosis
Keywords: Head Lice
MeSH Terms: conditions — Lice Infestations | interventions — Permethrin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Malathion Gel (Experimental): Malathion gel 0.5% 30 minute application
  Interventions: Drug: Malathion gel 0.5%
- Nix Crème Rinse (Active Comparator): Nix Crème Rinse applied to scalp for 10 minutes
  Interventions: Drug: Permethrin 1% rinse (Nix Crème)

INTERVENTIONS:
Drug: Malathion gel 0.5% — Malathion gel 0.5% applied to scalp for 30 minutes. May be repeated in 1 week if head lice are still present.
  Arms: Malathion Gel
Drug: Permethrin 1% rinse (Nix Crème) — Permethrin 1% shampooed into scalp for 10 minutes. May be repeated in 1 week if head head lice are still present.
  Arms: Nix Crème Rinse

SUMMARY:
In this study, Malathion Gel 0.5% will be compared to Nix (permethrin 1%) as a treatment for head lice in patients 2 years of age and older. Malathion Gel 0.5% is a new formulation of an established head lice treatment. The new formulation has been evaluated in 2 previous studies of patients 2 years of age and older.

DETAILED DESCRIPTION:
This is a Phase III, multi-center, investigator-blinded, two-arm, randomized, parallel group study, evaluating the safety and efficacy of a Malathion Gel, 0.5% formulation, manufactured by Taro. The objective is to show superiority of the novel product to an active control, Nix® Crème Rinse, manufactured by Insight Pharmaceuticals.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed active head lice infestation

Exclusion Criteria:

* Allergy to pediculicides or hair care products
* Scalp conditions other than head lice
* Previous head lice treatment within the past 4 weeks
* Current antibiotic treatment

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Investigator Site, Hot Springs, Arkansas
  - Investigator Site, Sacramento, California
  - Investigator Site, Kissimmee, Florida
  - Investigator Site, Miami, Florida
  - Investigator Site, Ormond Beach, Florida
  - Investigator Site, Picayune, Mississippi
  - Investigator Site, San Antonio, Texas

REFERENCES:
- [Result] Meinking TL, Vicaria M, Eyerdam DH, Villar ME, Reyna S, Suarez G. A randomized, investigator-blinded, time-ranging study of the comparative efficacy of 0.5% malathion gel versus Ovide Lotion (0.5% malathion) or Nix Creme Rinse (1% permethrin) used as labeled, for the treatment of head lice. Pediatr Dermatol. 2007 Jul-Aug;24(4):405-11. doi: 10.1111/j.1525-1470.2007.00460.x. PMID 17845167

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Malathion Gel | Nix Crème Rinse
Started | 206 | 197
Completed | 196 | 169
Not Completed | 10 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Malathion Gel | Nix Crème Rinse | Total
Number analyzed (Participants) | 206 | 197 | 403
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 161 | 154 | 315
  Between 18 and 65 years | 45 | 42 | 87
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.45 (11.81) [2 to 44] | 13.85 (12.80) [2 to 44] | 13.66 (12.30) [2 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 168 | 349
  Male | 25 | 29 | 54
Region of Enrollment [Number; unit: participants]
  United States | 206 | 197 | 403

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Index Subjects Free of Any Lice 14 Days After Their Last Treatment in the Modified ITT (LOCF)
Description: The primary efficacy variable was the proportion of index subjects who were considered a Treatment Success 14 days after their last treatment (Day 14 visit if only treated on Day 1, Day 21 visit if treated on Day 1 and Day 7)
  Treatment Success in the Efficacy ITT (LOCF)
  index subjects: 150 from 403 randomized (the youngest subject in the household that met the index case criteria (having nits and at least 3 live lice))
Time Frame: 3 weeks
Population: Efficacy: index subjects who had at least one application of treatment mITT: treated subjects who had at least one post-treatment visit Subjects with missing efficacy data were included first LOCF and then with non-LOCF PP: subjects who complied with the protocol, completed all required visits Safety: all subjects who had at least one treatment
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Crème Rinse
Number analyzed (Participants) | 75 | 75
percentage of subjects | 86.67 | 45.33
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Crème Rinse; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Proportion of Subjects Who Were Considered a Treatment Success 14 Days After Their First Treatment in the Modified ITT (LOCF).
Description: The secondary efficacy variable was the proportion of subjects who were considered a Treatment Success 14 days after their first treatment.
  Treatment Success in the Efficacy ITT (LOCF)
Time Frame: 3 weeks
Population: Proportion of subjects that are lice free 14 days after their first treatment
Measure: Number; unit: percentage of subjects
Arm/Group | Malathion Gel | Nix Crème Rinse
Number analyzed (Participants) | 198 | 184
percentage of subjects | 89.90 | 55.43
Statistical Analysis 1: Comparison: Malathion Gel vs Nix Crème Rinse; Test type: Superiority or Other; p = 0.0005, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Malathion Gel | Nix Crème Rinse
Serious Adverse Events (participants affected / at risk) | 0/206 | 0/197
Other Adverse Events (participants affected / at risk) | 21/206 | 37/197
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Malathion Gel (N=206) | Nix Crème Rinse (N=197)
APPLICATION SITE EROSION (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
APPLICATION SITE ERYTHEMA (Skin and subcutaneous tissue disorders) | 10 (11) | 5 (5)
APPLICATION SITE PRURITUS (Skin and subcutaneous tissue disorders) | 4 (4) | 19 (19)
APPLICATION SITE IRRITATION (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
CHEST DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CONJUNCTIVAL IRRITATION (Eye disorders) | 0 (0) | 3 (3)
EYE IRRITATION (Eye disorders) | 0 (0) | 1 (1)
INFLUENZA (General disorders) | 1 (1) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No